CLINICAL TRIAL: NCT06064760
Title: Values and Virtues of Grandparents Caring for Their Grandchildren as Protective Factors of Their Health and Psychological Wellbeing
Brief Title: Workshop on Strengths and Competences to Improve Psychological Wellbeing and Quality of Life of Grandparents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M02.0401.000.MPI20CNG
Record Dates: First submitted 2022-06-07; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-06

CONDITIONS: Psychological Well-being; Quality of Life; Virtues; Skill, Coping
Keywords: Grandparents-grandchildren relationship; Grandparents caregivers; Grandparenthood; Supplementary care; Psychological well-being; Quality of life; Personal strengths; Emotional competences; Psychoeducational group intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Quantitative, observational and longitudinal study with three measurements (pre-intervention, post-intervention and monitoring).
  The measurements will be taken before the intervention, at the end of the intervention and at three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group is given the Workshop on Strengths and Competences to Improve Psychological Wellbeing and Quality of Life of Grandparents.
  Interventions: Behavioral: Psychoeducational Workshop on Personal Strengths and Emotional Competences to Improve the Psychological Wellbeing and Quality of Life of Grandparents Caring for Their Grandchildren
- Control group (No Intervention): The control group is not given the Workshop on Strengths and Competences to Improve Psychological Wellbeing and Quality of Life of Grandparents.

INTERVENTIONS:
Behavioral: Psychoeducational Workshop on Personal Strengths and Emotional Competences to Improve the Psychological Wellbeing and Quality of Life of Grandparents Caring for Their Grandchildren — The intervention is a psychoeducational group workshop (6-8 participants). It includes 5 sessions of, approximately, 90 minutes. In addition, 3 months after the end of the workshop, a follow-up call will be organized with the participants. Due to the Covid-19 pandemic, the workshop will be held online.
  The sessions are:
  * Session 1: Defining my role as grandparent.
  * Session 2: Deepening my relationships.
  * Session 3: Growing as grandparent.
  * Session 4: Discovering my emotional world.
  * Session 5: Caring for others and caring for myself.
  Arms: Experimental group

SUMMARY:
Recent social and demographic changes in Western countries have led to a reorganization of the family relationships, such as grandparents-grandchildren bond. The Survey of Health, Ageing and Retirement in Europe (SHARE) shows, on the one hand, that 52% of grandparents are auxiliary caregivers of their grandchildren and, on the other hand, that more than 15% of grandparents regularly care for their grandchildren, being the Spanish percentage the second highest of Europe. Given these figures, it is clear that many grandparents today are playing an important role as socializing agents for their grandchildren.

According to this, grandparents play their socializing rol by passing on their grandchildren skills, experiences, values, beliefs and affection. This bond not only influences positively on grandchildren, but also on grandparents. Caring for grandchildren allows grandparents to resolve the crises of generativity and integrity of self, included in Erikson's Theory of Psychosocial Development. Moreover, high leves of generativity are related with greater personal growth, one of the dimensions of psychological wellbeing. However, the literature on the socializing rol of grandparents is scarce and has focus on the negative effects of caring for grandchildren. In contrast, recent studies demonstrates that caring for grandchildren has positive effect on grandparents' health and life satisfaction.

Being important to consider the negative consequences of this type of care, is also necessary to develop a new perspective, focus on protective factors of grandparents' psychological wellbeing and quality of life. According to McCubbin's Resilience Model of Family Stress, Adjustment and Adaptation, psychological resources and coping skills could be protective factors, minimizing the impact of caring for grandchildren.

The present project considers two protective factors: personal strengths and emotional competences, variables that are worked on the workshops. By focusing on these aspects, not only an improvement in family relationships (grandparents-parents-grandchildren) is expected, but also an increase in the psychological well-being and quality of life of the participants.

The development of intervention programs aimed at protective factors could be useful for grandparent caregivers, promoting their psychological well-being and quality of life.

DETAILED DESCRIPTION:
The study intervention consists of a psychoeducational group workshop oriented to grandparents caring for at least one minor grandchild.

The workshop includes 5 sessions and a follow-up call. The duration of the sessions is about 90 minutes. The modality is online.

The sessions and their objectives are detailed below:

- Session 1: Defining my role as a grandparent.

To frame the topic, get to know the participants and build a good group atmosphere.

- Session 2: Deepening my relationships.

To promote participants' confidence as grandparents.

- Session 3: Growing as a grandparent.

To help participants become aware of useful caregiving strategies.

- Session 4: Discovering my emotional world.

To help participants learn about and understand their own emotional world.

- Session 5. Caring for others and caring for me.

To help participants live their role as a grandparent without displacing other vital elements important to them.

- Follow-up. Phone call.

To offer participants a final one-on-one meeting.

ELIGIBILITY:
Inclusion Criteria:

* Being grandparent of, at least, one minor children or adolescent.

Exclusion Criteria:

* Suffer from a disease that makes the person unable to understand the questionnaire (e.g., moderate-severe dementia).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Grandparents' psychological wellbeing | Through study completion, an average of 2 years
  Psychological wellbeing will be evaluated with Ryff's Psychological Wellbeing Scale.
  Scale values: 1 (very inadequate to describe me), 2 (quite inadequate to describe me), 3 (some inadequate to describe me), 4 (some adequate to describe me), 5 (quite adequate to describe me), 6 (very adequate to describe me).
  Interpretation: the higher the score, the greater the psychological wellbeing of the person being assessed.
Grandparents' quality of life | Through study completion, an average of 2 years
  Quality of life will be evaluated with CASP-12.
  Scale values: 1 (sometimes), 2, 3, 4 (never).
  Interpretation: the higher the score, the greater the quality of life of the person being assessed.
Grandparents' involvement and burnout | Through study completion, an average of 2 years
  Involvement and burnout will be evaluated with Multidimensional Experience of Grandparenthood Set of Inventories.
  Scale values: 1 (totally disagree), 2, 3, 4, 5 (totally agree).
  Interpretation: the higher the score, the greater the involvement and burnout of the person being assessed as grandparent.
Grandparents' emotional competences | Through study completion, an average of 2 years
  Emotional competences will be evaluated with Grandparents Emotional Competency Scale.
  Scale values: 1 (never), 2 (sometimes), 3 (almost always), 4 (always).
  Interpretation: the higher the score, the greater the emotional competences of the person being assessed as grandparent.
Grandparents' character strengths | Through study completion, an average of 2 years
  Character strengths will be evaluated with Psychological Resources Inventory-77 items.
  Scale values: 0 (totally disagree), 1, 2, 3 (totally agree).
  Interpretation: the higher the score, the greater the character strengths of the person being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Noriega García, Principal Investigator — CEU San Pablo University
Locations (1):
- San Pablo CEU University (Campus Montepríncipe), Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in Excel format at https://osf.io/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from June 2023.
URL: http://osf.io/

REFERENCES:
- [Background] Arpino B, Bordone V, Balbo N. Grandparenting, education and subjective well-being of older Europeans. Eur J Ageing. 2018 Mar 20;15(3):251-263. doi: 10.1007/s10433-018-0467-2. eCollection 2018 Sep. PMID 30310372
- [Background] Chan, K. L., Chen, M., Lo, K. M. C., Chen, Q., Kelley, S. J., & Ip, P. (2018). The effectiveness of interventions for grandparents raising grandchildren: A meta-analysis. Research on Social Work Practice, 29(6), 1-11. https://doi.org/gf7j
- [Background] Diaz D, Rodriguez-Carvajal R, Blanco A, Moreno-Jimenez B, Gallardo I, Valle C, van Dierendonck D. [Spanish adaptation of the Psychological Well-Being Scales (PWBS)]. Psicothema. 2006 Aug;18(3):572-7. Spanish. PMID 17296089
- [Background] Erikson, E. H. (2000). El ciclo vital completado. Paidós.
- [Background] Findler, L., Taubman-Ben-Ari, O., Nuttman-Shwartz, O., & Lazar, R. (2013). Construction and validation of the multidimensional experience of grandparenthood set of inventories. Social Work Research, 37(3), 237-253. https://doi.org/10.1093/swr/svt025
- [Background] García, V., & Martínez-González, R. A (2017). Escala de competencias emocionales de abuelos y abuelas (ECEA). Revista Iberoamericana de Diagnóstico y Evaluación, 49(4), 107-120. https://doi.org/10.21865/RIDEP49.4.09
- [Background] Goodsell, T. L., Bates, J. S., & Behnke, A. O. (2011). Fatherhood stories: Grandparents, grandchildren, and gender differences. Journal of Social and Personal Relationships, 28, 134-154. https://doi.org/10.1177/0265407510386447
- [Background] Martínez de Serrano, B.A. (2007). Desarrollo y validación de un instrumento para la evaluación de los recursos psicológicos: Inventario de recursos psicológicos-77 ítems (IRP-77). Tesis doctoral publicada, Universidad Autónoma de Madrid, Madrid.
- [Background] McCubbin, M. A. (1993). Family stress theory and the development of nursing knowledge about family adaptation. In S. L. Feetham, S. B. Meister, J. M. Bell, & C. L. Gillis (eds.), The Nursing Family (pp. 46-58). Sage Publications.
- [Background] Moore SM, Rosenthal DA. Personal growth, grandmother engagement and satisfaction among non-custodial grandmothers. Aging Ment Health. 2015;19(2):136-43. doi: 10.1080/13607863.2014.920302. Epub 2014 Jun 9. PMID 24911594
- [Background] Noriega, C., Velasco, C., & López, J. (2020). Perceptions of grandparents' generativity and personal growth in supplementary care providers of middle-aged grandchildren. Journal of Social and Personal Relationships, 37, 1114-1135. https://doi.org/fvqh
- [Background] Park, N., Peterson, C., & Seligman, M. E. P. (2004). Strengths of character and well-being. Journal of Social and Clinical Psychology, 23(5), 603-619. https://doi.org/dg5xc7
- [Background] Perez-Rojo G, Martin N, Noriega C, Lopez J. Psychometric properties of the CASP-12 in a Spanish older community dwelling sample. Aging Ment Health. 2018 May;22(5):700-708. doi: 10.1080/13607863.2017.1292208. Epub 2017 Feb 28. PMID 28282724
- [Background] Peterson, C., & Seligman, M. E. P. (2004). Character strenghts and virtues. Oxford University Press. SHARE (29 de septiembre de 2021). La encuesta de salud, envejecimiento y jubilación en Europa. https://www.share.cemfi.es/index.asp?menu=1
- [Background] Sherr, L., Roberts, K. J., Hothi, S., & Balchin, N. (2018). Never too old to learn - parenting interventions for grandparents: A systematic review. Cogent Social Sciences, 4, 1-22. https://doi.org/10.1080/23311886.2018.1508627
- [Background] Triadó, C., Villar, F., Celdrán, M., & Solé, C. (2014) Grandparents who provide auxiliary care for their grandchildren: Satisfaction, difficulties, and impact on their health and well-being. Journal of Intergenerational Relationships, 12, 113-127. https://doi.org/10.1080/15350770.2014.901102
- [Background] Villar, F. (2012). Successful ageing and development: The contribution of generativity in older age. Ageing and Society, 32, 1087-1105. https://doi.org/fwpm7g
- [Background] Zhou J, Mao W, Lee Y, Chi I. The Impact of Caring for Grandchildren on Grandparents' Physical Health Outcomes: The Role of Intergenerational Support. Res Aging. 2017 Jun;39(5):612-634. doi: 10.1177/0164027515623332. Epub 2016 Jan 4. PMID 26733495

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT06064760/SAP_000.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT06064760/ICF_001.pdf